CLINICAL TRIAL: NCT02797496
Title: Comparison of Two Rehabilitation Programs in Patients With Mild to Moderate Parkinson's Disease. A Randomized, Controlled Study.
Brief Title: Comparison of Two Rehabilitation Programs in Patients With Mild to Moderate Parkinson's Disease.
Acronym: ASYMOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P071236; 2009-A00669-48 (Other: ID RCB)
Record Dates: First submitted 2016-06-08; First posted 2016-06-13 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Mild to moderate stage; Asymmetric Motor Strengthening; Rehabilitation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Asymmetric Motor Strengthening (Experimental)
  Interventions: Other: Asymmetric Motor Strengthening
- Conventional Therapy (Active Comparator)
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Other: Asymmetric Motor Strengthening — In the Asymmetric Motor Strengthening program, the principle is to concomitantly reinforce the "body openers" and stretch the "body closers". One alternates two types of practice during a session. Active exercises consist of fatiguing series of rapid alternating movements against light weights working on movements of extension/abduction/external rotation/supination. Stretch postures consists of short 1-2 minutes bouts of flexor/internal rotator/adductor/pronator stretch. The duration of rehabilitation program is 8 weeks.
  Arms: Asymmetric Motor Strengthening
Other: Conventional therapy — Conventional therapy will include general stretch, strengthening and balance exercises, respiratory exercises and relaxation methods.
  Arms: Conventional Therapy

SUMMARY:
Parkinson's disease is a major source of handicap, for which physical treatments are often underutilized with respect to chemical or surgical treatments. Yet, dopaminergic treatments alone prove unable to stop or control the gradual worsening of motor disability after a few years.

The training program that this study sets out to evaluate aims to restore balance between agonist extensors and antagonist flexors in Parkinson's disease.

There is indeed in Parkinson's disease an imbalance between weak flexors and weaker extensors, with excessive predominance of the flexors. The hypothesis of the study is that a motor strengthening program targeting extensor muscles specifically will improve body posture and restore motor function better than a conventional physical therapy program, in mild to moderate Parkinson's disease.

This is a parallel-group, single blind, randomized trial (investigators will be kept unaware of the physical treatment followed by study subjects).

The duration of patient participation is 5 months: 2-month intervention and 3-month follow-up following the intervention.

ELIGIBILITY:
Inclusion Criteria

* Patient diagnosed with Parkinson's disease on UKPDSBB criteria.
* Hoehn & Yahr stage 2, 3 in "OFF" state
* Age ≥18 years
* Patient who agreed to sign an informed consent to participate in this study.

Exclusion Criteria

* Patients who cannot or do not wish to follow a motor rehabilitation program for two months with a subsequent follow-up 3 months
* Intercurrent severe condition jeopardizing the vital or functional prognosis or the ability to participate in rehabilitation sessions.
* Cognitive dysfunction making effective communication or participation in a rehabilitation program impossible
* Person not benefiting from French State Health Insurance
* Current participation in another research protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-12; Primary Completion 2014-02 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in UPDRS (Unified Parkinson's Disease Rating Scale) III score in the " OFF " medication state, between baseline (D1) and Day 60 | Baseline (D1) and Day 60

SECONDARY OUTCOMES:
UPDRS III score in " ON " medication state | Baseline (Day 1), Day 60 and Day 150
UPDRS III score in " OFF " medication state | Day 150
Speed and step length over 20 meters (with 2 turn around, 2 Stand up-Sit down and 2 Sit down-Stand up) at maximal speed in " OFF " medication state | Day 1, Day 60 and Day 150
Motor power of neck, elbow and knee extensors, measured using a portable dynamometer at Day 1, Day 60 and Day 150 | Day 1, Day 60 and Day 150
Kinematic measurements of trunk inclination | Day 1 and Day 60
Balance measurement on posturography | Day 1 and Day 60
Quantitative testing of large vs small rapid alternating movement in the upper limbs (Hand Tapper) | Day 1, Day 60 and Day 150
Mount Sinai Parkinson Impairment Rating Scale | Day 1, Day 60 and Day 150
Global Mobility Task (GMT) | Day 1, Day 60 and Day 150
Geriatric Depression Scale - 15 items | Day 1, Day 60 and Day 150
Quality of life measured by PDQ-39 | Day 1, Day 60 and Day 150

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel GRACIES, Md, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

IPD SHARING:
Plan to Share IPD: Undecided